CLINICAL TRIAL: NCT00660855
Title: A Multicenter, Open Label Trial To Evaluate Analgesic Effect Of Intravenous And Subsequent Oral Therapy With Parecoxib/Valdecoxib (Bextra® IM/IV And Bextra®) 40 Mg/Day For Treatment Of Post-Laparoscopic Surgery Pain
Brief Title: A Multicenter, Open Label Trial To Evaluate Pain Relief With Intravenous Followed By Oral Therapy With Parecoxib/Valdecoxib 40 Mg/Day For Treatment Of Post-Laparoscopic Surgery Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See Detailed Description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3471107
Record Dates: First submitted 2008-04-01; First posted 2008-04-17 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Pain, Post Surgical
Keywords: laparoscopy
MeSH Terms: conditions — Pain, Postoperative | interventions — parecoxib; valdecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: parecoxib/valdecoxib

INTERVENTIONS:
Drug: parecoxib/valdecoxib — parecoxib 40 mg intravenously after recovery from anesthesia; if pain persisted, the patient could receive an optional second drug dose on Study Day 1 (only) if more than 4 hours after the first dose. When the patient was able to tolerate oral medication, one valdecoxib 40 mg tablet was administered by mouth once daily in the morning until a maximum period of 7 days.

SUMMARY:
The objectives of this study were to assess the analgesic efficacy and safety of parecoxib/valdecoxib on post-laparoscopic surgery analgesia.

DETAILED DESCRIPTION:
This study A3471107 was terminated on February 4th, 2005 due to enrollment difficulties, problems related to need for rescue medication, and perceptions about cardiovascular risk potentially associated with all NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone laparoscopic surgery
* Patients in need of post-surgical analgesia

Exclusion Criteria:

* Patients with an unexpected surgical complication which, in the Investigator's opinion, placed the patient at significantly higher risk for post-surgical complication(s), or for non-routine post-operative care requirements
* Patients who took any nonsteroidal anti-inflammatory drug or any analgesic within 48 hours prior to surgery

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-06; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale Pain Intensity (0-100 mm), which was evaluated using the change from baseline | Day 3

SECONDARY OUTCOMES:
Visual Analog Scale Pain Intensity | Day 7
Categorical Pain Intensity | Day 3 and Day 7
Patient pain relief | Day 3 and Day 7
Composite Upper Gastrointestinal (UGI) Tolerability measure was calculated; an UGI event was considered if the patient reported at least one of the following: moderate or severe nausea, or moderate or severe abdominal pain, or moderate or severe | Study endpoint
Dyspepsia | Study endpoint
Adverse events | Day 1, Day 3, and Day 7
Patient Global Evaluation | Day 3 and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Buenos Aires, Argentina

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3471107&StudyName=A%20Multicenter%2C%20Open%20Label%20Trial%20to%20evaluate%20pain%20relief%20with%20intravenous%20followed%20by%20oral%20therapy%20with%20parecoxib/valdecoxib%2040%20mg/day%20